CLINICAL TRIAL: NCT03079648
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Angelica Gigas N. Extract on Improvement of Blood Triglyceride
Brief Title: Efficacy and Safety of Angelica Gigas N. Extract on Improvement of Blood Triglyceride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WBP-HL-AG1
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Hyperlipidemias
Keywords: Angelica gigas N. extract; Hyperlipidemia; Clinical Trial
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angelica gigas N. extract (Experimental): capsules (2cap/d, 1,000mg/d) for 12 weeks.
  Interventions: Dietary Supplement: Angelica gigas N. extract
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Angelica gigas N. extract — capsules (2cap/d, 1,000mg/d) for 12 weeks.
  Arms: Angelica gigas N. extract
Dietary Supplement: Placebo — Placebo for 12 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Angelica gigas N. extract on improvement of Blood Triglyceride.

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. Twenty subjects were randomly divided into Angelica gigas N. extract or a placebo group. Fasting triglyceride profiles before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80 years with Triglyceride 130-200 mg/dL

Exclusion Criteria:

* Lipid lowering agent within past 6 months
* Severe cardiovascular disease(Mvocardial infarction, Stroke, etc)
* Renal disease(Heredity hyperlipidemia, Acute/Chronic renal failure, Nephrotic syndrome, etc)
* Cancer, Respiratory organ disease(Asthma, Chronic obstructive pulmonary disease)
* Autoimmune disease
* Diabetes mellitus
* Allergic or hypersensitive to any of the ingredients in the test products
* History of disease that could interfere with the test products or impede their absorption
* Under antipsychotic drugs therapy within past 2 months
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test by show the following results

  * aspartate aminotransferase, alanine aminotransferase > Reference range upper limit treble
  * Serum Creatinine > 2.0 mg/dl
* Pregnancy or breast feeding
* Not Contraception(except: Surgery for female infertility)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Changes of Triglyceride | 12 weeks
  Changes of triglyceride were assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of Lipid profile | 12 weeks
  Changes of Lipid profile were assessed before and after the intervention
Changes of Arteriosclerosis index | 12 weeks
  Changes of Arteriosclerosis index were assessed before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided